CLINICAL TRIAL: NCT02903667
Title: Biomaterial to Counteract Ridge Reduction Following the Removal of Multiple Adjacent Teeth. A Prospective Randomized Controlled Study.
Brief Title: Biomaterial to Counteract Ridge Reduction Following the Removal of Multiple Adjacent Teeth.
Acronym: Biomaterial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute Franci (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-2013-018
Record Dates: First submitted 2016-09-01; First posted 2016-09-16 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Alveolar Ridge Trauma; Bone Resorption
Keywords: bone grafting; implantology; oral surgery
MeSH Terms: conditions — Bone Resorption | interventions — Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bone grafting (Experimental): The possibility of counteracting unfavourable ridge modelling after multiple tooth extractions by placing bone grafting material in the fresh extraction sites.
  Interventions: Device: Bone grafting
- natural healing (Sham Comparator): ridge modelling after multiple tooth extractions.
  Interventions: Device: Bone grafting

INTERVENTIONS:
Device: Bone grafting

SUMMARY:
An open, prospective, randomized, multicenter study focused on the ridge diminution in case of grafting of fresh extraction sockets with Bio-Oss Collagen, Bio-Gide (Geistlich Pharma, Wolhusen, Switzerland), placing Dentsply implants (Astra Tech System).

DETAILED DESCRIPTION:
The removal of at least 2 adjacent teeth would cause more advanced hard tissue loss during healing than that occurring after removal of a single tooth with adjacent teeth present. In order to maintain the dimension of the ridge following tooth removal, bone grafts and bone substitutes have also been placed in the extraction socket. So far no data have been reported on the effect of removal of multiple adjacent teeth on bone loss at various aspects of the edentulous sites. Furthermore, the potential effect on ridge contraction of implant placement in multiple fresh extraction sites is not documented. Therefore, the objective of the study is to evaluate the possibility of counteracting un favourable ridge modeling after multiple tooth extractions by placing mineral bovine bone in the extraction sockets and covering the wound with a native collagen membrane. In addition, the possibility of placing implants in the grafted sites is evaluated after six month of healing. For these purpose 40 subjects with 2 or more fresh adjacent extraction sites in need of two or more implants replacing teeth will be enrolled. Ridge dimensional changes will be measured after 6 months of healing; marginal bone loss will be measured after 3-years follow-up from the baseline (prosthetic delivery).

ELIGIBILITY:
Inclusion Criteria:intact extraction sockets following removal of the natural teeth defined by:

* a marginal dehiscence defect of any of the facial bone walls of 3 mm
* no facial fenestration present in the apical of the marginal bone crest

Exclusion Criteria:

* untreated rampant caries and uncontrolled periodontal disease
* uncontrolled diabetes or any other systemic or local disease or condition that would compromise post-operative healing
* unable or unwilling to return for follow-up or unlikely to be able to comply with study procedures according to investigators judgement.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Cone Beam Computerized Tomographic (CBCT) examination at the center of each extraction socket, between the sockets, at the septum next to adjacent teeth. | Up to 24 weeks
  Measurements of alveolar ridge dimensional changes in the first 6 months of healing

SECONDARY OUTCOMES:
Standard intraoral radiograph of each experimental socket and inter-dental bone | 3 years follow up
  Changes in crestal bone level between baseline (prosthetic restoration) and follow-up (3 years later)

CONTACTS AND LOCATIONS:
Locations (1):
- Franci Institute, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided